CLINICAL TRIAL: NCT05844891
Title: Telehealth-Enhanced Asthma Care for Home After the Emergency Room (TEACH-ER)
Brief Title: Telehealth-Enhanced Asthma Care for Home After the Emergency Room
Acronym: TEACH-ER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sean Frey, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 00008286; R01HL169466 (NIH)
Record Dates: First submitted 2023-04-21; First posted 2023-05-06 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Research assistants conducting telephone follow-up assessments 3, 6, 9, and 12 months after enrollment will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth-Enhanced Asthma Care for Home After the Emergency Room (Experimental): New model of patient-centered asthma management.
  Interventions: Behavioral: Telehealth-Enhanced Asthma Care for Home After the Emergency Room (TEACH-ER)
- Enhanced Care (EC) Comparison Group (Active Comparator): Standard emergency department care for asthma exacerbations, enhanced through a report of recent symptoms sent to PCPs, and systematic feedback on asthma management/care at intervals that parallel the TEACH-ER group's telemedicine assessments.
  Interventions: Behavioral: Enhanced Care (EC)

INTERVENTIONS:
Behavioral: Telehealth-Enhanced Asthma Care for Home After the Emergency Room (TEACH-ER) — TEACH-ER aims to provide primary care management and educational support for families managing childhood asthma throughout the transition from emergency department to home, and includes several core components: 1) brief, pictorial, and health literacy-informed asthma education in the ED, with color- and shape-coded labels provided for home asthma medications; 2) virtual primary care follow-up within 1 week of discharge using in-home telemedicine (when possible), featuring provider prompts for guideline-based preventive therapy and home delivery of prescribed medications with pictorial action plans; 3) two additional in-home virtual visits to reinforce teaching, review treatment plans, label medications, and support effective management practices. Virtual visits will be completed using the Zoom platform on smartphones or other compatible devices. We anticipate that all three telehealth visits (1 provider visit, 2 educator visits) will be completed within 2 months of enrollment.
  Arms: Telehealth-Enhanced Asthma Care for Home After the Emergency Room
Behavioral: Enhanced Care (EC) — Similar to children in the TEACH-ER group, participants in the EC group will receive a symptom assessment using NHLBI guidelines, a recommendation for appropriate preventive medications, and asthma education materials given at the time of the ED visit. After baseline and randomization, we will send the child's PCP a symptom report with guideline-based recommendations for preventive care and recommend a follow-up visit with the PCP. We will also give all providers a summary of the current national guidelines. We will provide systematic feedback to the family and child's PCP at intervals that parallel the TEACH-ER group's telemedicine assessments. This feedback will include prompting caregivers to schedule a recommended follow-up appointment with the PCP, and encouraging providers to adhere to the NHLBI guidelines. While participants will not be blinded to their group allocation, they will be told that they are randomly assigned to two different ways of approaching asthma management.
  Arms: Enhanced Care (EC) Comparison Group

SUMMARY:
The investigators propose a randomized controlled trial of Telehealth-Enhanced Asthma Care for Home After the Emergency Room (TEACH-ER) vs. enhanced care (EC). TEACH-ER includes: 1) brief, pictorial, and health literacy-informed asthma education in the ED, with color- and shape-coded labels provided for home asthma medications; 2) virtual primary care follow-up within 1 week of discharge using in-home telemedicine (Zoom) when possible, featuring provider prompts for guideline-based preventive therapy and home delivery of prescribed medications with pictorial action plans; 3) two additional in-home virtual visits to reinforce teaching, review treatment plans, label medications, and support effective management practices. The investigators will enroll 430 children (ages 3-12 yrs) from the two dedicated pediatric EDs in our region, and follow all participants for a 12-month period. The investigators will call caregivers to complete blinded follow-up telephone surveys at 3, 6, 9, and 12 months after discharge. The investigators will assess the effectiveness of TEACH-ER in reducing the need for additional asthma-related ED visits or hospitalizations in the 1-months after enrollment. Additional outcomes of interest include asthma symptoms, medication adherence, absenteeism from work and school, quality of life, and the delivery of care consistent with national asthma care guidelines.

ELIGIBILITY:
Inclusion Criteria (all criteria must be met):

* Physician diagnosis of asthma, based on review of medical records and/or caregiver report.
* Current emergency visit for an acute asthma exacerbation, requiring treatment with rescue medication.
* Persistent asthma or poor asthma control for which a daily controller medication is recommended by NHLBI guidelines, defined as any 1 of the following:

  1. >2 days/wk with asthma symptoms in the past month,
  2. >2 days/wk with rescue medication use in the past month,
  3. >2 days/month with nighttime symptoms in the past month (vs. 1-2 nights per month if 3-4 years old), or
  4. ≥1 other episode of asthma during the past year that required systemic corticosteroids (vs. during the past 6 months if 3-4 years old).
* Child age between ≥3 and ≤12 years.
* Child and caregiver live in Monroe County, NY.

Exclusion Criteria:

* An inability to speak and understand English. Parents (and children) with low literacy / health-literacy skills will be eligible, as survey instruments will be administered verbally and educational materials will be designed for low-literacy populations.
* No access to a working phone for follow-up surveys (either at the subject's home or an easily accessible location). If a subject does not have access to an appropriate device for Zoom visits at home, we will provide a device with required data plan.
* Other significant medical conditions, including cystic fibrosis, congenital heart disease, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
* Children in foster care or other situations in which consent cannot be obtained from a legal guardian.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of asthma-related hospitalizations and emergency department visits after discharge | 12 months
  Asthma-related hospitalizations or emergency department visits, and drawn from objective healthcare utilization data in the electronic health record

SECONDARY OUTCOMES:
Symptom-Free Days (SFD) in the past 2 weeks | Baseline, 3 months, 6 months, 9 months, 12 months
  The number of 24-hour periods within the previous 14 days that a child remained free of asthma symptoms (range: 0-14 days); a higher score indicates more days without symptoms. Reported by caregivers during scheduled telephone assessments.
Caregiver-reported Asthma control (NHLBI) | Baseline, 3 months, 6 months, 9 months, 12 months
  Asthma control over the past 1 month, as based on caregiver report of recent symptoms, activity limitation, and medication use during scheduled telephone assessments.
Missed school due to asthma in the past 2 weeks | Baseline, 3 months, 6 months, 9 months, 12 months
  We will ask caregivers to report how many days of school the child missed (if any) during the previous 2 weeks due to their asthma (range: 0-14 days).
Missed work due to asthma in the past 2 weeks | Baseline, 3 months, 6 months, 9 months, 12 months
  We will ask caregivers to report how many days of work the caregiver missed (if any) during the previous 2 weeks due to their child's asthma (range: 0-14 days).
Caregiver-reported Medication adherence | Baseline, 3 months, 6 months, 9 months, 12 months
  Recent adherence with prescribed controller therapy as reported by caregivers during scheduled telephone assessments using the Medication Adherence Report Scale (5-25 points; higher scores indicate higher levels of reported adherence).
Caregiver quality of life | [Time Frame: 2 months, 4 months, 6 months]
  The Pediatric Asthma Caregiver Quality of Life Questionnaire (PACQLQ) is a well-established, validated measure of caregiver quality of life over the previous 1 week, as reported by caregivers during scheduled telephone assessments (score range: 1-7 points; 1 indicates severe impairment, 7 indicates no impairment).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No